CLINICAL TRIAL: NCT06038851
Title: Evaluation of the Analgesic Benefit of Adding the Blocks of the Intermediate and Medial Femoral Cutaneous Nerves in Addition to the Femoral Triangle Block for Postoperative Analgesia After a Knee Replacement Surgery: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Analgesic Benefit of Adding the Blocks of the Intermediate and Medial Femoral Cutaneous Nerves in Addition to the Femoral Triangle Block for Postoperative Analgesia After a Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23.116
Record Dates: First submitted 2023-08-29; First posted 2023-09-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Post-operative Pain; Anesthesia, Local
Keywords: total knee replacement surgery; para-sartorial compartments block; femoral triangle block
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Single-center, prospective superiority study, randomized controlled, triple blind
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Para-Sartorial Compartment (PACS) Block + Femoral Triangle Block (FTB) + IPACK block (Experimental): In addition to the injection performed in the femoral triangle, two injections of 5 mL of 0.5% ropivacaine + epi 1:400 000 will be performed below the sartorius muscle (subsartorial compartment) and above the sartorius muscle (suprasartorial compartment).
  For all patients, an infiltration between popliteal artery and capsule of the knee block (IPACK) will be performed concomitantly, in order to block the sensory branches of the innervation posterior to the knee with 15 ml of ropivacaine 0.3% + epi 1:400 000.
  Interventions: Procedure: Para-Sartorial Compartments (PACS) Block; Procedure: Femoral Triangle Block (FTB); Procedure: Infiltration between popliteal artery and capsule of the knee (IPACK) block
- Femoral Triangle Block (FTB) + IPACK block (Active Comparator): This block is currently the most used in practice and is considered a standard of care. It consists of a single injection of 15 ml of 0.5% ropivacaine + epi 1:400 000 under the sartorius muscle, lateral to the femoral artery, at the level of the apex of the femoral triangle
  For all patients, an infiltration between popliteal artery and capsule of the knee block (IPACK) will be performed concomitantly, in order to block the sensory branches of the innervation posterior to the knee with 15 ml of ropivacaine 0.3% + epi 1:400 000.
  Interventions: Procedure: Femoral Triangle Block (FTB); Procedure: Infiltration between popliteal artery and capsule of the knee (IPACK) block

INTERVENTIONS:
Procedure: Para-Sartorial Compartments (PACS) Block — This intervention was selected because it has the potential to optimize analgesia by skin coverage of the upper third of the surgical incision. The intervention will be performed as follows:
  * The intermediate femoral cutaneous nerve will be visualized at the supralateral level of the sartorius muscle, in a duplicature of the fascia lata.
  * The needle will be inserted at the same puncture site as for the femoral triangle block, with a latero-medial orientation in the plane (intracanalar compartment).
  * In addition to the injection performed in the femoral triangle, two injections of 5 mL of 0.5% ropivacaine + epi 1:400 000 will be performed in addition, below the sartorius muscle (subsartorial compartment) and above the sartorius muscle (suprasartorial compartment).
  Arms: Para-Sartorial Compartment (PACS) Block + Femoral Triangle Block (FTB) + IPACK block
Procedure: Femoral Triangle Block (FTB) — * The high frequency linear ultrasound probe will be positioned midway between the superior edge of the patella and the anterosuperior iliac spine. It will then be moved to visualize the apex of the femoral triangle, confirmed by visualization of the sartorius muscle laterally and the long adductor medially.
  * The needle will be inserted with a latero-medial orientation in the plane.
  * The initial injection will be a single injection of 15 ml of 0.5% ropivacaine + epi 1:400 000 under the sartorius muscle, lateral to the femoral artery, at the level of the apex of the femoral triangle.
Procedure: Infiltration between popliteal artery and capsule of the knee (IPACK) block — It will be performed in order to block the sensory branches of the innervation posterior to the knee with 15 ml of ropivacaine 0.3% + epi 1:400 000.

SUMMARY:
Total knee replacement surgery can be associated with a significant postoperative pain burden and an inability to mobilize adequately, which can lead to the failure of the ambulatory course.

Indeed, early mobilization is beneficial in this context in order to prevent complications related to immobility.

The optimization of postoperative analgesia is therefore a key issue for the success of this intervention in an outpatient setting or during a short-term hospitalization since an adequate pain relief facilitate the earlier mobilization of the operated joint. Modern postoperative analgesia protocols recommend a multimodal approach, including the use of acetaminophen, anti-inflammatories, opioids and others as well as the use of nerve blocks.

Some nerve blocks used for total knee replacement surgery, such as the femoral nerve block, do not preserve the motor skills of the operated limb, which may alter the clinical trajectory due to delayed mobilization due to weakening of the quadriceps, one of the extensor muscles of the knee. Currently, one of the blocks used to spare the motor functions is the block of the femoral triangle.

Unfortunately, this block of the femoral triangle does not fully cover the skin component of the surgical incision used for a total knee arthroplasty. A solution to obtain a better quality of pain relief at the level of the cutaneous incision would be to add a block of the para-sartorial compartment, which makes it possible to cover the nerve territories not covered by the femoral triangle block.

The hypothesis of this study is that the addition of the para-sartorial compartments (PACS) block, which aims to block the intermediate cutaneous femoral nerve, will improve the postoperative analgesia after total knee replacement surgery, compared to the classical isolated approach of the femoral triangle block (FTB).

DETAILED DESCRIPTION:
Despite many advances, the postoperative analgesia offered by the present techniques remains imperfect, the femoral triangle block does not make it possible to completely cover the cutaneous component of the classic midline incision used for a total knee arthroplasty. This incision would fall more under the anterior cutaneous femoral nerves, more specifically the intermediate and medial cutaneous femoral nerves. A recently described approach offers the prospect of better covering this skin incision, by specifically blocking these nerves using the same needle path as for the femoral triangle block. Although the feasibility of this approach has been studied in healthy volunteers and in a few clinical cases, no randomized controlled study has been conducted to determine whether the addition of cutaneous femoral nerve blocks offers an analgesic benefit in the population undergoing total knee replacement surgery. This is therefore necessary in order to assess whether this approach improves the clinical trajectory of patients receiving a total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over, requiring a primary total knee arthroplasty
* 'American Society of Anesthesiologists' classification 1 to 3

Exclusion Criteria:

* Refusal or unable to consent
* Contraindications to a peripheral nerve block;
* Inability to communicate with the healthcare team or the research team;
* Inability to understand follow-up instructions or questionnaires;
* Chronic pain requiring the intake of the equivalent of more than 60 mg of morphine daily;
* Pregnancy;
* Patients weighing less than 50 kg (to limit the risk of intoxication with local anesthetics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Intensity of the postoperative pain | 24 hours after the surgery
  The Pain Intensity short form questionnaire (PROMIS) is universal rather than disease-specific. The first two items in the Pain Intensity item bank assess pain intensity utilizing a 24-hour recall period (items include the phrase "the past 24 hours") while the last item asks patient to rate their pain intensity "right now."

SECONDARY OUTCOMES:
Intensity of the postoperative pain | 7 days after the surgery
  The Pain Intensity short form questionnaire (PROMIS) is universal rather than disease-specific. The first two items in the Pain Intensity item bank assess pain intensity utilizing a 7-day recall period (items include the phrase "the past 7 days") while the last item asks patient to rate their pain intensity "right now."
Total morphine consumption | 24 hours after the surgery
Time between the end of surgery and the first opioid dose | 24 hours after the surgery
Pain levels | 6 hours, 12 hours, 18 hours and 24 hours after the surgery
  Postoperative pain levels will be assessed every 6 hours for the first 24 hours after the surgery using a numerical scale where 0 = no pain and 10 = worst pain imaginable
Complications | 24 hours after the surgery
  The rate of complications or adverse effects during the first 24 hours will be assessed, such as local anesthetic toxicity, nausea, vomiting, pruritus and acute urinary retention.
Quality of sleep | 24 hours after the surgery
  The quality of sleep of the patient will be evaluated, rated on a scale where 0 = insomnia and 10 = excellent quality sleep.
Quality of postoperative recovery | Change between baseline (day 0) and 7 days after the surgery
  QoR15 is a valid questionnaire to measure the quality of recovery after surgery and anaesthesia, which includes 15 questions. Each of the 15 items are scored by the patient from 0 (worst score) to 10 (optimal score), giving a lowest possible score of 0 (worst outcome), and a highest possible score of 150 (optimal outcome).
Patient's satisfaction | 24 hours and 7 days after the surgery
  The satisfaction of the patient will be evaluated, rated on a scale where 0 = completely dissatisfied and 10 = fully satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Roy, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No